CLINICAL TRIAL: NCT05913739
Title: Impact of Oxygen Therapy on Readmissions of Patients With Chronic Heart Failure With Reduced Ejection Fraction
Brief Title: Oxygen Therapy in Patients With Chronic Heart Failure With Reduced Ejection Fraction
Acronym: ROXIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Marc Bonnin, MD, PhD. Marc Bonnin Vilaplana, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROXIC
Record Dates: First submitted 2023-02-08; First posted 2023-06-22 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Chronic Heart Failure; Oxygen Deficiency
Keywords: oxygen therapy
MeSH Terms: conditions — Hypoxia | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: A randomization of the patients will be carried out receiving oxygen therapy (treatment group) and those not receiving this treatment (control group): randomization will be done according to list
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen Therapy (Active Comparator): Participants received nocturnal oxygen therapy (minimum 6 hours) for 6 months.
  Interventions: Other: Oxygen Therapy
- No Oxygen Therapy (No Intervention): Participants will not received oxygen therapy

INTERVENTIONS:
Other: Oxygen Therapy — Nocturnal oxygen therapy minimum 6 hours
  Arms: Oxygen Therapy

SUMMARY:
The purpose of this study is to assess patients with chronic heart failure and moderate-severe ventricular dysfunction (left ventricular ejection fraction (FEVE) <40%) with nocturnal desaturation (mean Oxygen saturation (SatO2) <90% and/or Cummulative time (TC) <90% > 22 minutes) without underlying respiratory disease, oxygen treatment during hours of night rest will reduce exacerbations, improve the ability to effort, sleep quality and poor prognostic parameters of heart failure, compared to patients not receiving oxygen treatment.

DETAILED DESCRIPTION:
36 patients will attend at baseline, monthly, 3-month and 6-monthly visits.

BASELINE VISIT After being informed about the study and potential risks, all patients giving written informed consent, will be randomized (according to the list) receiving oxygen therapy (treatment group) and those not receiving this treatment (control group).

The following information will be collected:

* Demographics, pathological history, concomitant medication.
* Physical examination, vital signs (pressure, heart rate, weight)
* Doppler echocardiography (an echocardiography performed in the last 6 months will be accepted)
* Analytical determination of biomarkers NT-proBNP and ultrasensitive troponin.
* Assessment of baseline functional class by NYHA classification.
* Respiratory function tests: spirometry and diffusion (will accept tests performed in the last 6 months).
* Arterial blood gases.
* Nocturnal respiratory polygraphy.
* Exercise capacity with the 6-minute walk test (P6MM)
* Evaluation of health-related quality of life with the Minnesota questionnaire
* Assessment of sleep quality using the Pittsburgh questionnaire

If the patient belongs to the treatment group, the intervention will begin with oxygen therapy with a static concentrator and nasal cannula during the night at home, with a minimum compliance of six hours, following the usual clinical practice. Overnight pulse oximetry at home with oxygen will be performed to confirm if the prescribed flow rate is adequate to achieve a mean SatO2 >90% and/or that the correction of the CT90. If this is not achieved, it will be repeated, modifying the oxygen flow until the target is reached.

The control group will not undergo this intervention.

The rest of the medical treatment will be carried out according to the usual protocol of the Heart Failure Unit.

Follow up visits:

Clinical follow-up will be done at one month, three months and six months after the start of the intervention in the Chronic Respiratory Pathology Unit of Pneumology.

At 1 and 3 months

* Analytical determination of biomarkers nt-proBNP and ultrasensitive troponin (TnThs).
* Baseline functional class will be collected by New York Heart Association (NYHA) classification.
* Physical examination, vital signs (blood pressure (BP), Heart rate (HR), weight).
* Adverse effects and concomitant medication.

At 6 months

* Analytical determination of biomarkers nt-proBNP and ultrasensitive troponin (TnThs).
* Baseline functional class by NYHA classification will be collected.
* Physical examination, vital signs (BP, HR, weight).
* Evaluation of exercise capacity will be done by means of the 6-minute walk test (PM6M).
* Nocturnal pulse oximetry of control: treatment group with oxygen to evaluate the response and control group without oxygen to evaluate the evolution.
* Assessment of health-related quality of life with the Minnesota questionnaire.
* Sleep quality will be assessed using the Pittsburgh questionnaire.
* Adverse effects and concomitant medication.

In the follow-up periods (1, 3 and 6 months), the number of decompensations will be recorded:

* Hospitalizations for heart failure.
* Emergency care for heart failure requiring at least one dose of intravenous diuretic treatment.
* Need for outpatient intravenous depletive treatment due to the presence of congestive signs.

The study will be considered completed after 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old.
* Diagnosis and clinic of chronic heart failure with ventricular dysfunction with left ventricular ejection fraction (LVEF) <40% under optimal medical treatment regardless of its etiology and having presented at least one episode of decompensation (visits to the emergency room, hospitalizations and/or need for intravenous depletive treatment) during the last year.
* Nocturnal desaturation defined as mean SatO2 <90% and/or Cummulative time (TC) <90>22 minutes to nocturnal pulse oximetry done at home.
* Signed informed consent

Exclusion Criteria:

* Chronic lung disease (includes chronic obstructive pulmonary disease with Pulmonary respiratory function (PRF) (forced expiratory volume at one second/forced vital capacity (FEV1/FVC) <70%), diffuse interstitial diseases, pulmonary hypertension of respiratory).
* Obstructive sleep apnea-hypopnea syndrome (OSAHS) with Apnea hypopnea index (AHI) > 14.9.
* Previous treatment with oxygen therapy.
* Not agreeing to attend periodic cardiology visits.
* Being part of other clinical studies that contraindicate an intervention.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Nocturnal oxygen therapy at home in patients with heart failure heart rate and nocturnal desaturation can reduce the number of heart failure decompensations cardiac arrest. | changes from baseline to 6th month
  To assess whether treatment with nocturnal oxygen therapy at home in patients with heart failure heart rate and nocturnal desaturation (mean SatO2 <90% and/or CT <90%>22 minutes) no AOS manages to reduce the number of heart failure decompensations cardiac arrest (hospitalizations, visits to the emergency room or the need for depletive treatment intravenously) compared with patients not receiving oxygen therapy.

SECONDARY OUTCOMES:
Oxygen during the night rest is accompanied by reduction of the biomarker NTproBNP (pg/mL). Oxygen during the night rest is accompanied by reduction the biomarker TnThs (pg/mL). | changes from baseline to 6th month
  To analyze if the treatment with oxygen during the night rest is accompanied by reduction the biomarkers NTproBNP(pg/mL) and TnThs (pg/mL).
Nocturnal oxygen therapy on symptoms using the class function of the NYHA, in the capacity of effort (P6MM). | changes from baseline to 6th month
  To assess the benefit of nocturnal oxygen therapy on symptoms using the class function of the NYHA, in the capacity of effort (P6MM).
Nocturnal oxygen therapy on symptoms using the class function of the NYHA, in the quality of life (Minnesota score) | changes from baseline to 6th month
  To assess the benefit of nocturnal oxygen therapy on symptoms using the class function of the NYHA, in the quality of life (Minnesota score)
Nocturnal oxygen therapy on symptoms using the class function of the NYHA, in the quality of the dream (pittsburg score). | changes from baseline to 6th month
  To assess the benefit of nocturnal oxygen therapy on symptoms using the class function of the NYHA, in the quality of the dream (pittsburg score).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Girona Dr. Josep Trueta, Girona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) collected data can be shared as long as it is for research collaboration
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once the manuscript is accepted for publication
Access Criteria: Study data access will be provided for collaborative purposes

REFERENCES:
- [Background] Bekfani T, Abraham WT. Current and future developments in the field of central sleep apnoea. Europace. 2016 Aug;18(8):1123-34. doi: 10.1093/europace/euv435. Epub 2016 May 26. PMID 27234869
- [Background] Oldenburg O, Wellmann B, Buchholz A, Bitter T, Fox H, Thiem U, Horstkotte D, Wegscheider K. Nocturnal hypoxaemia is associated with increased mortality in stable heart failure patients. Eur Heart J. 2016 Jun 1;37(21):1695-703. doi: 10.1093/eurheartj/ehv624. Epub 2015 Nov 26. PMID 26612581
- [Background] Khayat R, Jarjoura D, Porter K, Sow A, Wannemacher J, Dohar R, Pleister A, Abraham WT. Sleep disordered breathing and post-discharge mortality in patients with acute heart failure. Eur Heart J. 2015 Jun 14;36(23):1463-9. doi: 10.1093/eurheartj/ehu522. Epub 2015 Jan 29. PMID 25636743
- [Background] Watanabe E, Kiyono K, Matsui S, Somers VK, Sano K, Hayano J, Ichikawa T, Kawai M, Harada M, Ozaki Y. Prognostic Importance of Novel Oxygen Desaturation Metrics in Patients With Heart Failure and Central Sleep Apnea. J Card Fail. 2017 Feb;23(2):131-137. doi: 10.1016/j.cardfail.2016.09.004. Epub 2016 Sep 9. PMID 27615064
- [Background] Gottlieb JD, Schwartz AR, Marshall J, Ouyang P, Kern L, Shetty V, Trois M, Punjabi NM, Brown C, Najjar SS, Gottlieb SS. Hypoxia, not the frequency of sleep apnea, induces acute hemodynamic stress in patients with chronic heart failure. J Am Coll Cardiol. 2009 Oct 27;54(18):1706-12. doi: 10.1016/j.jacc.2009.08.016. PMID 19850211
- [Background] Bradley TD, Logan AG, Kimoff RJ, Series F, Morrison D, Ferguson K, Belenkie I, Pfeifer M, Fleetham J, Hanly P, Smilovitch M, Tomlinson G, Floras JS; CANPAP Investigators. Continuous positive airway pressure for central sleep apnea and heart failure. N Engl J Med. 2005 Nov 10;353(19):2025-33. doi: 10.1056/NEJMoa051001. PMID 16282177
- [Background] Cowie MR, Woehrle H, Wegscheider K, Angermann C, d'Ortho MP, Erdmann E, Levy P, Simonds AK, Somers VK, Zannad F, Teschler H. Adaptive Servo-Ventilation for Central Sleep Apnea in Systolic Heart Failure. N Engl J Med. 2015 Sep 17;373(12):1095-105. doi: 10.1056/NEJMoa1506459. Epub 2015 Sep 1. PMID 26323938
- [Background] Damy T, Margarit L, Noroc A, Bodez D, Guendouz S, Boyer L, Drouot X, Lamine A, Paulino A, Rappeneau S, Stoica MH, Dubois-Rande JL, Adnot S, Hittinger L, d'Ortho MP. Prognostic impact of sleep-disordered breathing and its treatment with nocturnal ventilation for chronic heart failure. Eur J Heart Fail. 2012 Sep;14(9):1009-19. doi: 10.1093/eurjhf/hfs085. Epub 2012 Jun 22. PMID 22730336
- [Background] Yumino D, Bradley TD. Central sleep apnea and Cheyne-Stokes respiration. Proc Am Thorac Soc. 2008 Feb 15;5(2):226-36. doi: 10.1513/pats.200708-129MG. PMID 18250216
- [Background] Levi-Valensi P, Weitzenblum E, Rida Z, Aubry P, Braghiroli A, Donner C, Aprill M, Zielinski J, Wurtemberger G. Sleep-related oxygen desaturation and daytime pulmonary haemodynamics in COPD patients. Eur Respir J. 1992 Mar;5(3):301-7. PMID 1572442
- [Background] Toyama T, Seki R, Kasama S, Isobe N, Sakurai S, Adachi H, Hoshizaki H, Oshima S, Taniguchi K. Effectiveness of nocturnal home oxygen therapy to improve exercise capacity, cardiac function and cardiac sympathetic nerve activity in patients with chronic heart failure and central sleep apnea. Circ J. 2009 Feb;73(2):299-304. doi: 10.1253/circj.cj-07-0297. Epub 2008 Dec 27. PMID 19122308
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Shigemitsu M, Nishio K, Kusuyama T, Itoh S, Konno N, Katagiri T. Nocturnal oxygen therapy prevents progress of congestive heart failure with central sleep apnea. Int J Cardiol. 2007 Feb 14;115(3):354-60. doi: 10.1016/j.ijcard.2006.03.018. Epub 2006 Jun 23. PMID 16806535
- [Background] du Bois RM, Weycker D, Albera C, Bradford WZ, Costabel U, Kartashov A, King TE Jr, Lancaster L, Noble PW, Sahn SA, Thomeer M, Valeyre D, Wells AU. Forced vital capacity in patients with idiopathic pulmonary fibrosis: test properties and minimal clinically important difference. Am J Respir Crit Care Med. 2011 Dec 15;184(12):1382-9. doi: 10.1164/rccm.201105-0840OC. Epub 2011 Sep 22. PMID 21940789
- [Background] Yi H, Shin K, Shin C. Development of the sleep quality scale. J Sleep Res. 2006 Sep;15(3):309-16. doi: 10.1111/j.1365-2869.2006.00544.x. PMID 16911033
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Background] Julious, S.A. Sample size of 12 per group rule of thumb for a pilot study. .Pharmaceutical Statistics. 2005; 4: 287-291.
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081